CLINICAL TRIAL: NCT02375399
Title: New Approaches to Echocardiography Assessment of Cardiac Dyssynchrony: Relevance Concerning Response Rate to Cardiac Resynchronization Therapy
Brief Title: New Echocardiographic Parameters for Prediction of Response to Cardiac Resynchronization Therapy
Acronym: NEW-CRT
Status: Terminated | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Mathias Konstandin, M.D., Heidelberg University
Other Study IDs: S-553/2012
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Echocardiography parameters for cardiac dyssynchrony had no predictive value in current multicentric prospective studies concerning cardiac resynchronization therapy. Comprehensive echocardiography and new parameters as 2D and 3D strain, as well as 3D echo have been analyzed, but their definite value has not been proven yet.

DETAILED DESCRIPTION:
In patients with severe heart failure, delays in the conduction system can result in asynchronous contraction impairing cardiac function. By implantation of pacemaker systems with three leads located in atrium, right ventricle and coronary sinus, tracing back this deranged contraction closer to the physiological excitation propagation is aimed (cardial resynchronization therapy [CRT]). Despite patient selection according to the guidelines nearly one-third of the patients do not profit, neither clinically nor echocardiographically, from an implanted CRT-device. In addition, recent studies have shown that no reliable prediction may be achieved with the known echocardiographic parameters of dyssynchrony, regarding the response to such therapy. The aim of this study is therefore to assess new echocardiographic parameters, which may allow to better predict CRT response.

ELIGIBILITY:
Inclusion Criteria:

* congestive heart failure, dilated cardiomyopathy, indication for implantation of a CRT-device according to the European Society of Cardiology (ESC)

Exclusion Criteria:

* persons who are incapable of giving informed consent
* acute heart attack
* arrhythmia during the examination (such as atrial fibrillation and frequent VES)
* state after STEMI with an extended scar
* inotropic drug therapy
* pre-existing permanent pacemaker stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred to the University Hospital of Heidelberg with congestive heart failure to undergo the implantation of CRT device
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
3D echocardiography | 12 months
  offline analysis of echocardiography data
2D strain | 12 months
  offline analysis of echocardiography data
m-mode echocardiography | 12 months
  offline analysis of echocardiography data

SECONDARY OUTCOMES:
NYHA | 12 months
  New York Heart Association (NYHA) functional classification
six-min walk test | 12 months
  distance walked over 6 minutes as a sub-maximal test of aerobic capacity
NT-proBNP | 12 months
  N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
LV EF | 12 month
  left ventricular (LV) ejection fraction (EF)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Konstandin, M.D., Principal Investigator — Heidelberg University
Locations (1):
- Department of Cardiology, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany